CLINICAL TRIAL: NCT01113450
Title: Results of a Program of Newborn Hearing Screening in Cuiaba-Brazil
Brief Title: Results of a Program of Newborn Hearing Screening (NHS) in Cuiaba-Brazil
Status: Completed | Type: Observational
Sponsor: Centro de Diagnostico Auditivo de Cuiaba (Other)
Responsible Party: Priscila de Araujo Lucas Rodrigues, CEDAC
Other Study IDs: TAN Cuiaba
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2009-12

CONDITIONS: Showing the Results of a Program of NHS in Cuiaba_ Brazil
Keywords: hearing, newborn, screening

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims to demonstrate the indices of quality of a Newborn Hearing Screening (NHS).

DETAILED DESCRIPTION:
The data refer to infants underwent newborn hearing screening by evoked otoacoustic emissions by transient stimulation, using the analyzer EOA Biologic. Examinations archived in the computer's service were analyzed for the amount of infants who passed or failed the screening, as well as the correlations with the same age and gender.

ELIGIBILITY:
Inclusion Criteria:

* middle ear conditions integrates

Exclusion Criteria:

* middle ear conditions inadequate

Ages: 2 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: There were two groups:
  1. high risk for hearing loss
  2. low risk for hearing loss
Sampling Method: Non-Probability Sample
Enrollment: 3148 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscila L Rodrigues, PHD student, Principal Investigator — Centro de Diagnostico Auditivo de Cuiaba
Locations (1):
- CEDAC, Cuiabá, Mato Grosso, Brazil